CLINICAL TRIAL: NCT06609590
Title: A Comparative Study Between Ultrasound Guided Anterior Glenoid Block Combined With Sub-omohyoid Anterior Suprascapular Block Versus Ultrasound Guided Interscalene Block in Diagnostic Shoulder Arthroscopy
Brief Title: A Comparative Study Between Anterior Glenoid Block With Sub-omohyoid Suprascapular Block Versus Interscalene Block in Shoulder Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, riham fathy galal, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FAMSU R143/2024
Record Dates: First submitted 2024-09-14; First posted 2024-09-24 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients will receive Anterior glenoid block combined with suprascapular nerve block.
  Interventions: Procedure: Glenoid nerve block combined with Sub-omohyoid Anterior Suprascapular nerve Block
- Group B (Experimental): The patients will Interscalene brachial plexus block.
  Interventions: Procedure: Interscalene brachial plexus block

INTERVENTIONS:
Procedure: Glenoid nerve block combined with Sub-omohyoid Anterior Suprascapular nerve Block — Ultrasound guided anterior glenoid nerve block combined with Sub-omohyoid Anterior Suprascapular nerve Block
  Arms: Group A
Procedure: Interscalene brachial plexus block — Ultrasound guided interscalene brachial plexus block
  Arms: Group B

SUMMARY:
The patients will be randomized into 2 equal groups by a computer-generated random numbers table, named group A, B.

Group A: Patients will receive Anterior glenoid block combined with suprascapular nerve block.

Group B: Patients will receive conventional interscalene block.

In group A, the patient will be supine for anterior glenoid block.

The suprascapular nerve will be identified as it branch off from the superior trunk and will be traced until it courses beneath the inferior belly of the omohyoid muscle.

In group B, interscalene brachial plexus block will be performed.

The primary outcomes will be as follows: (1) 11-point (0-10) numeric rating scale (NRS) pain score immediately before surgery starts and after surgery; (2) degree of preserved diaphragmatic function (DPDF): the ratio of postoperative to pre-block (baseline) diaphragmatic excursion amplitude will be assessed in the holding area using a curvilinear probe (Sono Site, Transportable fuji M-turbo ultrasound system).;(3) degree of preserved handgrip strength (DPHS): the ratio of postoperative to pre-block (baseline) handgrip strength (the maximal force patients exerted when instructed to squeeze the dynamometer handles as tightly as feasible). Measurements will be done before surgery, immediately postoperative, 4, 8, and 24 hours postoperatively.

And (4) Recording of the complications which are: Hematoma, nerve injury, allergy to any of the used drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients American Society of anesthesiologists' physical status (ASA) I to II.
2. Aged 18 to 65 years.
3. Both sexes.
4. Patients scheduled for shoulder arthroscopy.

Exclusion Criteria:

1. Patient refusal
2. ASA physical status III or more.
3. Patients with known allergy to any of the study drugs.
4. Infection at the site of injection.
5. Patients with history of cardiovascular disease.
6. Patients with renal disease.
7. Patients with hepatic disease.
8. Patients with neuromuscular disease.
9. Presence of any coagulopathy.
10. Chronic opioid, gabapentin or pregabalin use.
11. Patients with history of any psychiatric disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Degree of preserved diaphragmatic function (DPDF) | 24 hours postoperative.
  degree of preserved diaphragmatic function (DPDF): the ratio of postoperative to pre-block (baseline) diaphragmatic excursion amplitude will be assessed in the holding area using a curvilinear probe (Sono Site, Transportable fuji M-turbo ultrasound system).). Measurements will be made before surgery, immediately postoperative, 4, 8, and 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No